CLINICAL TRIAL: NCT06671925
Title: Targeting Loneliness in the Context of Chronic Pain Self-Management: An Intervention for Older Adults Living in Rural Areas
Brief Title: A Community Health Worker-Led Program for Chronic Pain and Loneliness in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Northern Michigan Health Consortium (Unknown); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary Janevic, Research Associate Professor Department of Health Behavior and Health Equity University of Michigan School of Public Health, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00261437; P30AG022845 (NIH)
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCOOP Intervention Group (Experimental): SCOOP is a 7-week intervention, delivered primarily over the telephone by community health workers, to support chronic pain self-management and social connectedness.
  Interventions: Behavioral: Strengthening COnnections to Overcome Pain (SCOOP)
- Control group (No Intervention): Control group participants receive usual care between the baseline and 8-week follow-up survey. After completing the follow-up survey, control participants will be invited to take part in an educational workshop about pain and loneliness and will receive all intervention materials.

INTERVENTIONS:
Behavioral: Strengthening COnnections to Overcome Pain (SCOOP) — Each week for 7 weeks, SCOOP intervention group participants will watch a brief video on the study website teaching a pain management or social connectedness skill and have a session with a community health worker, where they will receive support with behavioral goal-setting related to pain management and/or social connections. Participants will be screened for unmet social needs and connected to appropriate resources.
  Arms: SCOOP Intervention Group

SUMMARY:
The goal of this clinical trial is to test a new community health worker-delivered program (Strengthening COnnections to Overcome Pain, or SCOOP) that teaches strategies for managing chronic pain and loneliness to older adults living in rural areas. The main questions it aims to answer are:

1. Does participating in SCOOP result in less pain interference with daily life?
2. Does participating in SCOOP result in decreased loneliness?
3. What is the level of participant engagement in SCOOP? Researchers will compare people who have participated in SCOOP with people who have not participated in SCOOP to see if SCOOP is helpful in decreasing pain interference and loneliness.

Participants will:

1. Watch brief videos teaching strategies to manage pain and boost social connections.
2. Engage in up to 7 weekly coaching sessions with a community health worker.
3. Complete two telephone interviews about health, mental health, and functioning: one at baseline, and one 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 60 years;
* Have a mobile or landline phone;
* Self-reported chronic musculoskeletal pain (pain in muscles or joints for >= 3 months, >=4 (0-10 scale) average pain level over last week, >=1 day/previous 30 when pain made it difficult to do usual activities);
* Self-reported loneliness (Feeling lonely "some of the time" or more often);
* Able to converse comfortably in English.

Exclusion Criteria:

* Serious acute illness or hospitalization in the last month;
* Planned major surgery in the next three months that would interfere with program participation (e.g., knee or hip replacement);
* Severe cognitive impairment or other severe physical or psychiatric disorder judged by study team to pose a significant barrier to participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Engagement as measured by number of sessions completed | 8 weeks from baseline
  Number of sessions out of 7 that participants have completed 8 weeks from baseline.

SECONDARY OUTCOMES:
Participant satisfaction with the SCOOP intervention | 8 weeks from baseline
  Items ask about overall satisfaction with the program, i.e., whether participation increased understanding of pain management and increased knowledge of strategies to improve social connection (1= Strongly Disagree to 5= Strongly Agree). The mean of the two items will be calculated. A higher score indicates greater participant satisfaction with the intervention.
Change in Loneliness as measured by the UCLA 8-item Loneliness Scale | Baseline, 8 weeks from baseline
  Eight items ask about feelings of loneliness and social isolation. Each question is rated on a 4-point scale: 1=never, 2=rarely, 3=sometimes, and 4 =always. Two positively worded items ("I am an outgoing person" and "I can find companionship when I want it" are reverse-scored. All items are summed to give a total score of 8 to 32 points. A higher score indicates a greater degree of loneliness.
Change in Pain Interference 6-item subscale from PROMIS-43 Adult Profile | Baseline, 8 weeks from baseline
  Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference). Scores are converted to a standardized T-score metric, with a mean of 50 and a standard deviation of 10 in a referent population. A higher score means more of the concept being measured.

OTHER OUTCOMES:
Global Impression of Change in Pain, Functioning, and Loneliness | 8 weeks from baseline
  Three items, analyzed separately: 1) How participant thinks their pain has changed from baseline (much worse (-3) to much better(+3)). 2) How participant thinks their functioning has changed from baseline (much worse (-3) to much better(+3)). 3) How participant thinks their feelings of loneliness have changed from baseline (much worse (-3) to much better(+3)).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States